CLINICAL TRIAL: NCT01847989
Title: A Randomized, Placebo-controlled Single-dose, Double-blind Study of the Safety and Pharmacokinetics of Recombinant Factor XIII in Healthy Volunteers
Brief Title: Safety and Pharmacokinetics of Recombinant Factor XIII in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: F13-1661
Record Dates: First submitted 2013-05-02; First posted 2013-05-07 (Estimated); Last update posted 2017-01-11 (Estimated); Status verified 2017-01

CONDITIONS: Congenital Bleeding Disorder; Congenital FXIII Deficiency; Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- rFXIII (Experimental)
  Interventions: Drug: catridecacog
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: catridecacog — Single doses of rFXIII administered intravenously (IV) to eight subjects in each of the five dose groups (2, 5, 10, 25 and 50 U/kg).
  Arms: rFXIII
Drug: placebo — Single doses of placebo administered intravenously (IV) to two subjects in each of the five dose groups (2, 5, 10, 25 and 50 U/kg).
  Arms: Placebo

SUMMARY:
This trial was conducted in Europe. The aim of this trial was to investigate safety and pharmacokinetics of escalating single doses of catridecacog (recombinant factor XIII, rFXIII) in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Normal platelet count and clotting parameters
* Adequate renal and hepatic function
* If female and of child-bearing potential, negative serum pregnancy test within 21 days of enrollment and a negative urine pregnancy test on admission to the clinical research unit
* If a sexually active male or a sexually active female of child-bearing potential,agreement to use a medically accepted form of contraception from the time of enrollment to completion of all follow-up study visits
* Negative drug and alcohol screens

Exclusion Criteria:

* Known antibodies or hypersensitivity to FXIII
* Known bleeding or hematologic disorder
* Known allergy to yeast
* Receipt of blood products within 30 days of screening
* Donation of blood within 30 days prior to enrollment
* Any surgical procedure in the 30 days prior to enrollment
* Previous history of autoimmune disorders involving autoantibodies, e.g., systemic lupus erythematosus
* Receipt of treatment with any experimental agent within 30 days of study enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2003-01; Primary Completion 2003-05 (Actual); Study Completion 2003-05 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Days 0-28

SECONDARY OUTCOMES:
Incidence of clinically significant changes from baseline in physical examination or laboratory measurements | Days 0-28
Incidence of rFXIII antibodies, as measured by ELISA (Enzyme-Linked Immuno Sorbent Assay) | Days 0-28
Incidence of yeast antibodies | Days 0-28

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Novo Nordisk Investigational Site, Berkshire, United Kingdom

REFERENCES:
- [Result] Visich JE, Zuckerman LA, Butine MD, Gunewardena KA, Wild R, Morton KM, Reynolds TC. Safety and pharmacokinetics of recombinant factor XIII in healthy volunteers: a randomized, placebo-controlled, double-blind, multi-dose study. Thromb Haemost. 2005 Oct;94(4):802-7. doi: 10.1160/TH05-04-0292. PMID 16270634
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com